CLINICAL TRIAL: NCT04173702
Title: The Effect of Different Support Surface on Postural Sway and Limits of Stability in Healthy Individuals
Brief Title: The Effect of Different Support Surfaces on Balance in Healthy Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Recep Tayyip Erdogan University Training and Research Hospital (Other)
Collaborators: Hacettepe University (Other)
Responsible Party: Principal Investigator, Melek Merve ERDEM, Research Assistant, Recep Tayyip Erdogan University Training and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: GO 19/86
Record Dates: First submitted 2019-05-06; First posted 2019-11-22 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Healthy
Keywords: Balance; Stance width; Postural sway; Limits of stability

STUDY DESIGN:
Intervention Model Description: Clinical trials with a single arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy Group (Experimental): Postural sway and stability limits in assessment of healthy individuals
  Interventions: Diagnostic Test: balance analysis

INTERVENTIONS:
Diagnostic Test: balance analysis — Computerized balance analysis system will use to evaluate postural sway and limits of stability at four different support surfaces.

SUMMARY:
This study will evaluate how age, visual sensation and different ground properties affect of postural sways and stability limits at different support surface widths. 60 individuals will be included in this study.

DETAILED DESCRIPTION:
Balance is considered to be an important component of performance during activity as a result of a complex process in which musculoskeletal and neurological systems function. Two different balance states are defined as the static balance where the individuals maintain their inactive position or the dynamic balance when they perform a foreseen movement. The balance is maintained by keeping the center of gravity within the boundaries of the support surface and is provided by sensory impulses from the visual, vestibular and somatosensory systems organized by the central nervous system. Balance is an important factor to lead an independent life, and it is imperative that the balance be ensured in order to ensure that daily living activities are performed safely. The neural control of the bipedal posture varies depending on the width of the supporting surface, which has a significant impact on the frontal plane biomechanics. There is a linear relationship between increased support surface size and mechanical stability. In experimental studies, it has been shown that increasing muscle width levels in response to translational perturbations seen on the support surface on the horizontal plane have decreased with increasing step width. The changes in the preferred support surface vary depending on the age of the external environment, recurrent falls due to decreased sensory input, or various neurological disorders. However, there are few quantitative studies examining the relationship between different support surface widths and equilibrium, and the effect of posture width on sensory feedback control is still poorly understood. This study was planned to evaluate the effect of age, visual sensation and different soil properties on postural release and stability limits at different support surface widths.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals aged between 18-50
* Without any diagnosed disease
* Individuals who voluntarily agree to participate in this research

Exclusion Criteria:

* The presence of previous lower extremity surgery
* Pain during evaluation
* Foot ankle instability
* Important and irreversible visual deficits
* Body mass index (BMI) greater than> 40 kg / m²
* Limitation of ankle, knee and hip joint in lower extremity
* Muscle strength of the lower extremity (dorsiflexors, plantar flexors, quadriceps, hamstring, gluteus maximus, gluteus medius) and the trunk (rectus abdominous, internal and external oblique abdominals, back extensor) below 5.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-01-17 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-10-16 (Actual)

PRIMARY OUTCOMES:
Postural Sway | 1 week
  Postural sways were used to evaluate dynamic balance. Postural sway, in terms of human sense of balance, refers to horizontal movement around the center of gravity. Postural sway was assessed during quite standing with open/closed eyes on a hard/soft floor with the Bertec Balance System on 4 different support surfaces: adjacent feet, width of the bitrochanteric diameter, increased by 50% width of the bitrochanteric diameter and reduced by 50% of the width of the bitrochanteric diameter randomly.

SECONDARY OUTCOMES:
The Limits of Stability | 1 week
  The limits of stability were used to evaluate static balance. Limits of stability is the greatest distance in any direction a person can lean away from a midline vertical position without falling, stepping, or reaching for support. Participants were assessed with a force platform (Model BP 5050; Bertec Corporation, Columbus, Ohio) in terms of support surfaces on limits of stability (LoS) in the right, left, front and back directions when the eyes were open on the hard floor with the Bertec Balance System on 4 different support surfaces: adjacent feet, width of the bitrochanteric diameter, increased by 50% width of the bitrochanteric diameter and reduced by 50% of the width of the bitrochanteric diameter randomly.

CONTACTS AND LOCATIONS:
Overall Officials: Melek M. ERDEM, Principal Investigator — Tayyip Erdogan University Training and Research Hospital; Semra TOPUZ, Assoc. Prof., Study Director — Hacettepe University; Ozden OZKAL, PT, PhD, Study Chair — Hacettepe University; Ali I. Yalcin, PT, M.Sc., Study Chair — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Altindag, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, CSR
Time Frame: Data will be available within 6 months with completion of the result report.
Access Criteria: Requestors will be required to sign a Data Access Agreement.
URL: https://orcid.org/0000-0003-4073-3084

REFERENCES:
- [Background] Goodworth AD, Mellodge P, Peterka RJ. Stance width changes how sensory feedback is used for multisegmental balance control. J Neurophysiol. 2014 Aug 1;112(3):525-42. doi: 10.1152/jn.00490.2013. Epub 2014 Apr 23. PMID 24760788